CLINICAL TRIAL: NCT07268170
Title: Heart Rate Control: Betablockers or Ivabradine Therapy Before Cardiac Computed Tomography
Brief Title: Heart Rate Control Before Cardiac Computed Tomography in Adults for the Evaluation of Coronary Artery Disease
Acronym: HEART-BEAT
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-522741-21-00; 2025-522741-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Coronary Arterial Disease (CAD); Ischemic Heart Disease (IHD)
Keywords: Cardiac computed tomography; premedication; metoprolol; ivabradine; atenolol; heart rate control; heart rate
MeSH Terms: conditions — Myocardial Ischemia | interventions — Atenolol; Metoprolol; Ivabradine

STUDY DESIGN:
Intervention Model Description: Initial dose-finding pilot study using a controlled, double-blind, 6 armed 1:1 randomized design.
  Followed by a sequential controlled, double-blind, placebo-controlled study of most effective betablocker and ivabradine dose among a subgroup of diabetics and non-diabetics undergoing cardiac computed tomography.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Metoprololtartrat 50 mg (Experimental): Strategy 1
  Interventions: Drug: atenolol; Drug: Ivabradine
- Metoprololtartrat 100 mg (Experimental): Strategy 1
  Interventions: Drug: atenolol; Drug: Ivabradine
- Atenolol 50 mg (Experimental): Strategy 1
  Interventions: Drug: Metoprolol tartrate; Drug: Ivabradine
- Atenolol 100 mg (Experimental): Strategy 1
  Interventions: Drug: Metoprolol tartrate; Drug: Ivabradine
- Ivabradine 15 mg (Experimental): Strategy 1
  Interventions: Drug: atenolol; Drug: Metoprolol tartrate
- Ivabradine 7.5 mg (Experimental): Strategy 1
  Interventions: Drug: atenolol; Drug: Metoprolol tartrate
- Fastest dose of betablocker (atenolol 50/100 mg or metoprololtartrat 50/100 mg) (Experimental): Strategy 2
  Interventions: Drug: Ivabradine 7.5/15 mg
- Fastest dose of Ivabradine (Ivabradine 7.5/15 mg) (Experimental): Strategy 2
  Interventions: Drug: Atenolol/Metoprolol tartrate
- Placebo (Placebo Comparator): Strategy 2
  Interventions: Drug: Atenolol/Metoprolol tartrate; Drug: Ivabradine 7.5/15 mg

INTERVENTIONS:
Drug: atenolol — No studies have compared metoprololtartrat, ivabradine, atenolol and placebo in different doses as drugs before cardiac computed tomography
  Arms: Ivabradine 15 mg; Ivabradine 7.5 mg; Metoprololtartrat 100 mg; Metoprololtartrat 50 mg
Drug: Metoprolol tartrate — No studies have compared metoprololtartrat, ivabradine, atenolol and placebo in different doses as drugs before cardiac computed tomography
  Arms: Atenolol 100 mg; Atenolol 50 mg; Ivabradine 15 mg; Ivabradine 7.5 mg
Drug: Ivabradine — No studies have compared metoprololtartrat, ivabradine, atenolol and placebo in different doses as drugs before cardiac computed tomography
  Arms: Atenolol 100 mg; Atenolol 50 mg; Metoprololtartrat 100 mg; Metoprololtartrat 50 mg
Drug: Atenolol/Metoprolol tartrate — No studies have compared metoprololtartrat, ivabradine, atenolol and placebo in different doses as drugs before cardiac computed tomography
  Arms: Fastest dose of Ivabradine (Ivabradine 7.5/15 mg); Placebo
Drug: Ivabradine 7.5/15 mg — No studies have compared metoprololtartrat, ivabradine, atenolol and placebo in different doses as drugs before cardiac computed tomography
  Arms: Fastest dose of betablocker (atenolol 50/100 mg or metoprololtartrat 50/100 mg); Placebo

SUMMARY:
The goal of this clinical trial is to describe which type and dose of commonly used heart rate reducing drugs (metoprolol, atenolol, or ivabradine) has the swiftest heart rate reduction from baseline in patients aged 30 to 80 years with a heart rate > 65 beats per minute undergoing cardiac computed tomography for the evaluation of coronary artery disease. The main question it aims to answer is

• Which type of heart reducing drug and dose has the swiftest heart rate reduction before cardiac computed tomography?

DETAILED DESCRIPTION:
This single-center, prospective, randomized, double-blind, clinical trial will include patients undergoing cardiac computed tomography. Two phases will be conducted: a pilot study (dose-finding phase) and a randomized trial (superiority phase). In the first dose-finding phase participants (N=150) will be randomized 1:1 in six arms (arms contain lower and higher doses of atenolol, metoprolol and ivabradine). Following an interim analysis, a superiority phase will be conducted using two parallel groups, non-diabetics (N=100) and diabetics (N=100), in a placebo-controlled head-to-head randomized 2:2:1 three-arms trial comparing the fastest betablocker and dose and the fastest dose of ivabradine from the dose-finding phase.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are to undergo Cardiac CT
* Sinus rhythm with heart rate > 65 bpm on ECG
* Competent patients who have given written informed consent

Exclusion Criteria:

* Age > 80 years
* Age < 30 years
* Heart rate > 100 bpm
* BMI > 35
* Previous percutaneous coronary intervention (with or without stent)
* Previous CABG
* Known ischemic heart disease
* Pacemaker
* Acute coronary syndrome
* Known allergy to beta-blockers
* Known allergy to ivabradine
* Known allergy to used radiographic contrast agents
* Pregnant, including potentially pregnant, or breastfeeding (potentially pregnant patients will undergo pregnancy testing)
* Heart failure with systolic left ventricular ejection fraction < 45%
* Reduced kidney function with estimated glomerular filtration rate (eGFR) < 40 ml/min
* Regular treatment with beta-blockers
* Regular treatment with ivabradine
* Regular treatment with non-dihydropyridine calcium antagonists (Verapamil and Diltiazem)
* Regular treatment with Cordarone
* Contraindications for beta-blockers or ivabradine:
* Severe asthma
* Severe COPD
* Sick sinus syndrome
* Sinoatrial block (1st degree AV block)
* Advanced AV block (2nd or 3rd degree)
* Hypotension (systolic blood pressure < 110 mmHg)
* Severe heart failure
* Severe restrictive cardiomyopathy
* Severe aortic stenosis
* Severe circulatory disturbances
* Severe metabolic conditions
* Untreated pheochromocytoma
* Concurrent treatment with potent inhibitors of CYP3A4
* Concurrent treatment with potent inhibitors of MAO inhibitors,
* Concurrent treatment with potent inhibitors of CYP2D6 inhibitors
* Concurrent treatment with potent inhibitors of intravenous calcium antagonists type I or III

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose and type of drugs with the swiftest heart rate reduction in patients undergoing cardiac computed tomography | From adminstration of study drug to start af cardiac computed tomography, 2 hours
  Time in minutes to heart rate (mean) lowered by 10% from baseline after administration of study drug

SECONDARY OUTCOMES:
Proportion of patients with heart rate <60 beats per minute | From adminstration of study drug to start af cardiac computed tomography, 2 hours
Total heart rate reduction in beats per minute after 120 minutes | From adminstration of study drug to start af cardiac computed tomography, 2 hours
Number of patients in need of an intravenous betablocker | From adminstration of study drug to start af cardiac computed tomography, 2 hours
  Patients with a heart rate >60 beats per minutes after 2 hours after administration of study drug
Efficacy of intravenous administration of betablocker | From adminstration of study drug to start af cardiac computed tomography, 2 hours
  How patients tolerate intravenous betablocker
Evaluation of side effects, safety, and tolerability of metoprolol, atenolol, and ivabradine | From intervention af study drug to phone contact to patient 1 week after cardiac computed tomography
  Phone contact to patient to describe any side effects and the tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Morten Böttcher, Professor, Study Chair — University Clinic of Ishemic Heart Disease, Gødstrup Hospital; Simon Winther, MD, PhD, Principal Investigator — University Clinic of Ishemic Heart Disease, Gødstrup Hospital
Locations (1):
- University Clinic of Ischemic Heart Disease, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. All data will be analyzed and managed locally at our site, and we do not plan to share IPD.